CLINICAL TRIAL: NCT02681640
Title: Phase II Trial: uPAR PET/CT for Preoperative Staging of Breast Cancer Patients
Brief Title: uPAR PET/CT for Preoperative Staging of Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Curasight ApS (Unknown)
Responsible Party: Principal Investigator, Dorthe Skovgaard, MD, PhD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CS-2015-1
Record Dates: First submitted 2016-02-04; First posted 2016-02-12 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- uPAR PET (Experimental): One injection of 68Ga-NOTA-AE105 followed by Positron Emission Tomography (PET/CT scan) to evaluate possible axillary lymph node metastatic lesions
  Interventions: Other: 68Ga-NOTA-AE105; Device: Positron Emission Tomography PET/CT

INTERVENTIONS:
Other: 68Ga-NOTA-AE105 — One injection of 68Ga-NOTA-AE105
Device: Positron Emission Tomography PET/CT — Following injection of 68Ga-NOTA-AE105 the patients will be subjected to Positron Emission Tomography PET/CT

SUMMARY:
The sensitivity and specificity of uPAR PET/CT for preoperative detection of lymph node metastases in breast cancer.

DETAILED DESCRIPTION:
The sensitivity and specificity of uPAR PET/CT for detection of lymph node metastases will be tested by observer-blinded readings (two separate teams) and compared to diagnostic performance of conventional preoperative diagnostic workup procedures. The reference test will be histopathology of lymph nodes obtained by operative lymph node dissection (SN/ALND). Primary end point dichotomized: +/- lymph node metastases in ipsilateral axilla.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-verified breast cancer
* Primary tumor more than 2 cm (ultrasound or clinically)
* The participants must be capable of understanding and giving full informed written consent

Exclusion Criteria:

* Pregnancy
* Lactation/breast feeding
* Weight above 140 kg
* Treatment with neoadjuvant chemotherapy
* Known allergy towards the IMP

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03; Primary Completion 2017-02-10 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of uPAR PET/CT in identifying axillary lymph node metastases from breast cancer | 1 hour
  Two separate teams of certified specialists (1 radiology and 1 nuclear medicine) will based on uPAR-PET/CT assess the presence of metastases in axillary lymph nodes ("spread"/"no spread"). Lymph Node sampling and histopathology determine true positives and true negatives.

SECONDARY OUTCOMES:
Number of axillary lymph node metastasis | 1 hour
  Two separate teams of certified specialists (1 radiology and 1 nuclear medicine) will based on uPAR-PET/CT assess the number of metastases in axillary lymph nodes. Lymph node sampling and histopathology determine true positives and true negatives.
Number of distant metastases | 1 hour
  Two separate teams of certified specialists (1 radiology and 1 nuclear medicine) will based on uPAR-PET/CT assess the number of distant metastases. Biopsy/follow up imaging will be used as reference.

OTHER OUTCOMES:
Optimal time point for performing PET/CT following injection of 68Ga-NOTA-AE105 | 0-60 minutes
  The first 5 patients will be subjected to 60 minutes of dynamic PET imaging covering the breast tumor area, starting at the time of injection. The PET scan will be divided into 12 time frames of each 5 minutes. The time frame with the best visual tumor to background contrast, will be designated as the optimal time point p.i. for uPAR-PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe Skovgaard, MD PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No